CLINICAL TRIAL: NCT00581880
Title: Measuring Hope and Hopelessness in Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Fordham University (Other); Calvary Hospital, Bronx, NY (Other); Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: William Breitbart, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 04-145
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2009-01-15 (Estimated); Status verified 2009-01

CONDITIONS: Advanced Cancer
Keywords: end stage; Terminally Ill
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Terminally Ill patients
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires — A battery of questionnaires concerning your thoughts, opinions, and attitudes about your illness and outlook on life. In addition, we will ask to provide some background information about you and your illness. The questions will take approximately 30 to 45 minutes to complete. You fill out the questionnaire once only.

SUMMARY:
The purpose of this study is to develop an accurate and useful way of measuring patients' thoughts and feelings about hope and hopelessness as they relate to their illness. Doctors and psychologists from Memorial Sloan-Kettering Cancer Center, Calvary Hospital, the Peter MacCallum Cancer Centre, and Fordham University are working together to design a new measure. Findings from this research will help us study the nature of illness and develop improved methods of diagnosis and treatment. We hope what we learn from you will help us learn more about how to care better for patients with cancer and other severe illnesses.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Patients who are able to understand verbal and written English.
* Diagnosis of cancer.
* Patients with advanced cancer receiving ambulatory or inpatient care at Memorial Sloan-Kettering Cancer Center in New York City. Patients at Calvary Hospital and Peter MacCallum Cancer Centre admitted for palliative care will also be eligible for participation in this study

Exclusion Criteria:

* The presence of a psychotic mental disorder (e.g., Bipolar Disorder, Schizophrenia, Schizo-affective illness, psychosis due to substance abuse) as indicated in medical chart.
* Cognitive impairment so severe (i.e., Mini-Mental State exam score of less than 20) that, in the opinion of the Principal Investigator or Project Coordinator, would interfere with a patient's ability to give informed consent for research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited in equal numbers from Memorial Hospital and Calvary Hospital or Peter MacCallum Cancer Centre at each stage of data collection.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2005-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To explore and better understand the construct of hopelessness as it applies to terminally ill cancer patients. | conclusion of study
To develop a brief self-report measure of hopelessness grounded in the construct of hopelessness as it applies to terminally ill cancer patients. | conclusion of study

SECONDARY OUTCOMES:
To establish the reliability and validity of this newly developed measure of hopelessness in a large sample of terminally ill cancer patients. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: William Breitbart, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org